CLINICAL TRIAL: NCT04360811
Title: Assessment of Obstetric, Fetal and Neonatal Risks and Vertical SARS-CoV-2 Transmission During COVID-19 Pandemic by Creation and Analysis of a Biological and Tissue Collection of Pregnancy Outcomes
Brief Title: Assessment of Obstetric, Fetal and Neonatal Risks and Vertical SARS-CoV-2 Transmission During COVID-19 Pandemic
Acronym: COroFet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RC31/20/0123
Record Dates: First submitted 2020-04-22; First posted 2020-04-24 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Pregnancy
Keywords: Pregnant women; pandemic; COVID-19; vertical mother-fetal transmission; SARS-CoV-2
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Unexposed group : COVID 19 negatif pregant woman (Other): COVID-19 negative women (not immunize
  Interventions: Diagnostic Test: COVID 19 diagnostic test by PCR
- Exposed group : COVID 19 positif pregant woman (Other): Women positive for COVID-19 (symptomatic and asymptomatic) COVID-19 negative women with long-standing immunity
  Interventions: Diagnostic Test: COVID 19 diagnostic test by PCR

INTERVENTIONS:
Diagnostic Test: COVID 19 diagnostic test by PCR — 1. Inclusion of patients with clinical data (in a eCRF) and various samples collection according to the outcome of pregnancy
  2. Storage and freezing samples for subsequent analysis by RT-PCR COVID-19 (maternal saliva, cord blood, fetal stools, placenta, fetal tissue, amniotic fluid according to pregnancy outcomes) and by maternal and newborn and / or fetal serologies testing
  3. Pathological study of placentas and fetal autopsies
     * Histology of positive COVID-19 placentas
     * Brain and visceral histology of positive COVID-19 fetuses autopsied
  4. Analysis of patient comorbidities and comparison in the different groups
  5. Final statistical analysis

SUMMARY:
A new coronavirus (COVID-19) highlighted at the end of 2019 in China is spreading across all continents. Most often at the origin of a mild infectious syndrome, associating benign symptoms (such as fever, cough, and headache) to different degrees, COVID-19 can cause serious pulmonary pathologies and sometimes death. Data on the consequences during pregnancy are limited. The first Chinese data published seem to show that the symptoms in pregnant women are the same as those of the general population. There are no cases of intrauterine maternal-fetal transmission, but cases of newborns infected early suggest that there could be vertical intrauterine, perpartum or neonatal transmission. Prematurity and cases of respiratory distress in newborns of infected mothers have been described. Subsequently, an in-depth analysis of cases in pregnant women and pregnancy issues are necessary in order to improve knowledge on the subject.

DETAILED DESCRIPTION:
The main objective of this project is to set up a biological and tissue collection in order to study the transplacental passage of the SARS-CoV-2 virus, and the pregnancy outcomes (miscarriage, intra uterine fetal death, medical termination of pregnancy or living birth) during COVID-19 pandemic. The biological and tissue collection will be made up of systematic samples taken from parturient women and their pregnancy outcome at the time of their arrival at the maternity unit to deliver whatever their term and pregnancy outcome. This inclusion will concern all pregnant women, both symptomatic and asymptomatic positive COVID-19 women, and negative COVID-19 women. All women included will have a serological test to check their immunity status to SARS-CoV-2 in order to study pregnant women with an unnoticed COVID-19 infection during their pregnancy. The inclusion time will extend from the epidemic period until a year after, in order to document the outcomes of pregnant women potentially exposed to SARS-CoV-2 in early pregnancy. Samples analyses will be carried out after the epidemic peak to not overload laboratories in times of crisis.

The challenge is to have a better knowledge of the SARS-CoV-2 epidemiological and virological characteristics in particular its involvement in maternal-fetal morbidity and mortality, and to better understand the organs affected and the pathways of contamination within this particular mother-child duo.

ELIGIBILITY:
Inclusion Criteria:

* Women over 18 years old on the date of inclusion
* Pregnant women coming to deliver in the Paule de Viguier maternity unit of Toulouse's University Hospital between April 2020 and April 2021 regardless the pregnancy outcomes (live births, IUFD, miscarriages, medical termination of pregnancy ) and the term
* Women affiliated to a social security system (including AME)

Exclusion Criteria:

* Voluntary termination of pregnancy
* Language barrier
* Patient under a legal protection measure (guardianship, curatorship, or safeguard of justice)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 2494 (Actual)
Dates: Start 2020-04-17 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
number of positive COVID-19 women | Day 0
  Exposure to SARS-CoV-2 will be measured the day of delivery by RT-PCR on maternal saliva and by serology on maternal blood

SECONDARY OUTCOMES:
number of positive COVID-19 women | Day 0
  Description of the number of positive COVID-19 RT-PCRs in the conception products: amniotic fluid, frozen placenta fragment, frozen fetal tissue, cord blood or frozen cord fragment

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Dubucs, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital of Toulouse, Toulouse, France